CLINICAL TRIAL: NCT01778582
Title: Perspective-taking, and Examining the Clinical Trial Informed Consent Process
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913021; 13-C-N021
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2015-09-18

CONDITIONS: Emotions; Informed Consent
Keywords: Emotion; Informed Consent

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- Very few people with cancer participate in clinical trials. Some are uncertain about the treatment, or are afraid of being treated like a guinea pig. They may also feel that they have inadequate information about the trial. One possible way of encouraging people to sign up for clinical trials is to improve the informed consent process. Researchers want to understand how people read and understand informed consent documents.

Objectives:

- To study perspective taking, and to study how people understand the information and enrollment process for a clinical trial.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* This study will require one study visit.
* Participants will watch one of four movie clips. They will be asked to respond to the film by looking at it from the main character s perspective. They will then answer questions about how the clips made them feel.
* Participants will read a sample cancer clinical trial consent form on a computer. The computer will record their eye movements while they read the text. They will then be asked whether they remember the information in the consent form, and whether they would participate in the trial.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
This study aims to examine perspective-taking and emotional states. The study also aims to examine information processing in the context of clinical trial consent forms, perceptions of risk of study side effects, hypothetical intentions to enroll, and satisfaction with the consent review process. Adult human subjects will be randomly assigned to watch a movie and take the main character s. Participants will also be asked to read a consent form for a clinical trial. Finally, they will be asked a series of questions about the consent form. I have also attached changes to the lay summary, which I had previously submitted, just to make sure that you have them.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Participants who are currently being treated for cancer will be excluded because their experience of a cancer clinical trial consent form would be qualitatively different from a noncancer patient s experience. Similarly, because individuals who have participated previously in a clinical trial might have a different perspective on participation or let previous experienced bias their perceptions of the hypothetical clinical trial context, we will also exclude individuals who have previously participated in a medical clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11-15; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-08 (Actual)

PRIMARY OUTCOMES:
Assess knowledge of side effects to participate in a clinical trial | 1 year
Assess knowledge of risk perceptions to participate in a clinical trial | 1 year
Assess knowledge of hypothetical intentions to participate in a clinical trial | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Ferrer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Angie AD, Connelly S, Waples EP, Kligyte V. The influence of discrete emotions on judgement and decision-making: a meta-analytic review. Cogn Emot. 2011 Dec;25(8):1393-422. doi: 10.1080/02699931.2010.550751. Epub 2011 May 24. PMID 21500048
- [Background] Appelbaum PS, Roth LH, Lidz CW, Benson P, Winslade W. False hopes and best data: consent to research and the therapeutic misconception. Hastings Cent Rep. 1987 Apr;17(2):20-4. PMID 3294743
- [Background] Arora A, Rajagopalan S, Shafiq N, Pandhi P, Bhalla A, Dhibar DP, Malhotra S. Development of tool for the assessment of comprehension of informed consent form in healthy volunteers participating in first-in-human studies. Contemp Clin Trials. 2011 Nov;32(6):814-7. doi: 10.1016/j.cct.2011.05.012. Epub 2011 Jun 1. PMID 21664491